CLINICAL TRIAL: NCT07044544
Title: A Phase I Trial to Evaluate the Safety and Efficacy of Addition of Novel Anti-leukemia Agents to Flu/Mel RIC Transplant for High-risk Myeloid Malignancies
Brief Title: Trial of Novel Anti-leukemia Agents in Flu/Mel RIC Transplant for Myeloid Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Omer Jamy, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014728 (UAB 2469); Robert Award (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Myeloid Malignancy; Hematologic Malignancy; Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Leukemia; allogeneic transplant
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Granulocyte Colony-Stimulating Factor; Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: G-CSF + Decitabine (100mg/m2 bid for 2d) (Experimental): Cohort 1 DL1: G-CSF + Decitabine (100mg/m2 bid for 2d)
  G-CSF will be administered subcutaneously on days -14 to -10 at a dose of 5mcg/kg. Hold for wbc >20k.
  Decitabine will be investigated at two dose levels. 100mg/m2 bid for 2 days at dose level 1 and 50mg/m2 bid for 2 days at dose level -1. It will be administered as IV in days -11 and -10.
  Interventions: Drug: G-CSF; Drug: Decitabine
- Cohort 1 DL-1: G-CSF + Decitabine (50mg/m2 bid for 2d) (Experimental): Cohort 1 DL-1: G-CSF + Decitabine (50mg/m2 bid for 2d)
  G-CSF will be administered subcutaneously on days -14 to -10 at a dose of 5mcg/kg. Hold for wbc >20k.
  Decitabine will be investigated at two dose levels. 100mg/m2 bid for 2 days at dose level 1 and 50mg/m2 bid for 2 days at dose level -1. It will be administered as IV in days -11 and -10.
  Interventions: Drug: G-CSF; Drug: Decitabine
- Cohort 2: G-CSF + Decitabine + Ven (200mg/d for 7d) (Experimental): Cohort 2 DL1: G-CSF + Decitabine + Ven (200mg/d for 7d)
  G-CSF will be administered subcutaneously on days -14 to -10 at a dose of 5mcg/kg. Hold for wbc >20k.
  Decitabine will be investigated at two dose levels. 100mg/m2 bid for 2 days at dose level 1 and 50mg/m2 bid for 2 days at dose level -1. It will be administered as IV in days -11 and -10.
  Venetoclax will be investigated at two dose levels. 200mg daily for 7 days as dose level 1 of cohort 2 of the study and 400mg daily for 7 days as dose level 2. It will be administered orally on from days -12 to -6.
  Venetoclax 400 and 200 mg/day dose will be adjusted if the patient was on fluconazole (down to 200 and 100 mg/day), posaconazole or isavuconazole (100 and 50 mg/day), and voriconazole (50 and 25 mg/day)
  If cohort 2 DL1 clears the DLT period based on the criteria discussed previously, then we will start accruing patients to DL2 of cohort 2.
  Interventions: Drug: G-CSF; Drug: Decitabine; Drug: Venetoclax
- Cohort 2 DL2: G-CSF + Decitabine + Ven (400mg/d for 7d) (Experimental): Cohort 2 DL2: G-CSF + Decitabine + Ven (400mg/d for 7d)
  G-CSF will be administered subcutaneously on days -14 to -10 at a dose of 5mcg/kg. Hold for wbc >20k.
  Decitabine will be investigated at two dose levels. 100mg/m2 bid for 2 days at dose level 1 and 50mg/m2 bid for 2 days at dose level -1. It will be administered as IV in days -11 and -10.
  Venetoclax will be investigated at two dose levels. 200mg daily for 7 days as dose level 1 of cohort 2 of the study and 400mg daily for 7 days as dose level 2. It will be administered orally on from days -12 to -6.
  Venetoclax 400 and 200 mg/day dose will be adjusted if the patient was on fluconazole (down to 200 and 100 mg/day), posaconazole or isavuconazole (100 and 50 mg/day), and voriconazole (50 and 25 mg/day)
  Interventions: Drug: G-CSF; Drug: Decitabine; Drug: Venetoclax

INTERVENTIONS:
Drug: G-CSF — Granulocyte colony-stimulating factor (G-CSF) is a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream.
Drug: Decitabine — Decitabine is a hypomethylating agent.
  Other Names: Dacogen
Drug: Venetoclax — Venetoclax is a selective inhibitor of BCL-2 protein.
  Arms: Cohort 2 DL2: G-CSF + Decitabine + Ven (400mg/d for 7d); Cohort 2: G-CSF + Decitabine + Ven (200mg/d for 7d)

SUMMARY:
The purpose of this study is to determine the safety of adding Decitabine and Venetoclax to patients undergoing reduced intensity allogenic transplantation for treatment of hematologic malignances with Fludarabine and Melphalan.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability and preliminary activity of decitabine and venetoclax as part of RIC AHSCT in patients with high-risk AML and MDS. The study will follow a standard 3+3 design commonly used in phase I studies. Dose-adjustments will be made based on the incidence of dose-limiting toxicities (DLTs). The DLT period is from the first dose of decitabine to day 28 post-transplant.

Cohort 1 DL1: G-CSF + Decitabine (100mg/m2 bid for 2d) Cohort 1 DL-1: G-CSF + Decitabine (50mg/m2 bid for 2d) Cohort 2 DL1: G-CSF + Decitabine + Ven (200mg/d for 7d) Cohort 2 DL2: G-CSF + Decitabine + Ven (400mg/d for 7d)

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, age 18-75 years
2. Patients must have a related or unrelated peripheral blood stem cell donor. Sibling donor must be a 6/6 match for HLA-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing, and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation. Unrelated donor must the following: have Optimum: HLA-A, -B, -C, -DRB1, -DRB3/4/5, -DQA1, -DQB1, -DPA1 and -DPB1; Minimum: HLA-A, -B, -C, -and DRB1 matching at high resolution using DNA-based typing and be willing to donate peripheral blood stem cells and be medically eligible to donate stem cells according to National Marrow Donor Program (NMDP) criteria.
3. A candidate for reduced intensity preparative regimen, based on age≥60, or HCT-CI of ≥4, or considered by the treating physician to have high risk for toxicity with myeloablative preparative regimen.
4. Cardiac function: Ejection fraction >40%
5. Calculated creatinine clearance greater than 50 mL/minute (using the Cockcroft-Gault formula and actual body weight).
6. Pulmonary function: DLCO ≥50% (adjusted for hemoglobin) and FEV1≥50%
7. Liver function: total bilirubin < 1.5x the upper limit of normal and ALT/AST < 2.5x the upper normal limit. Patients who have been diagnosed with Gilbert's Disease are allowed to exceed the defined bilirubin value up to <3mg/dl.
8. Female subjects (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two effective methods of contraception or agree to complete abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.
9. Male subjects (even if surgically sterilized), of partners of women of childbearing potential must agree to practice effective barrier contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.
10. Karnofsky performance status KPS ≥ 70 (Appendix B)
11. Patients must have a diagnosis of one of the following:

    -AML: A. Any AML with active disease (defined as ≥ 5% blasts in the marrow), with no available re-induction strategies, or further therapy is not felt to be effective by treating physician.

    B. Any AML with adverse risk disease, therapy-related or secondary-AML in CR1 or beyond C. AML with intermediate risk disease that is MRD+ in CR1 or beyond D. Any AML in CR2 or beyond (regardless of MRD) E. Marrow blast percentage needs to be 20-25% and total WBC counts needs to be ≤ 25000/µl before the start of the conditioning regimen. It is acceptable to use hydroxyurea or low dose cytarabine to maintain this WBC count.

    -MDS:

    MDS with IPSS-M ≥ high and/or with ≥5% blasts in the bone marrow with no available pre-transplant strategies, or further therapy is not felt to be effective by treating physician.- MDS/MPN:

    -MDS/MPN >5% blasts and spleen < 22 cm with no available pre-transplant strategies, or further therapy is not felt to be effective by treating physician.
12. Subject is willing and able to sign informed consent and abide by the protocol requirements.

Exclusion Criteria:

1. Autologous hematopoietic stem cell transplant < 3 months prior to enrollment.
2. Previous allogeneic stem cell transplant.
3. Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
4. Known hypersensitivity to Decitabine, Venetoclax and/or ATG.)
5. Pregnant and/or breastfeeding
6. Evidence of HIV infection or known HIV positive serology.
7. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
8. Non-hematologic malignancy within prior three (3) years, with the exception of squamous cell or basal cell skin carcinoma. Patients with prior malignancies except resected localized non-melanoma skin cancer or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed as long as it is in remission. Cancer treated with curative intent < 5 years previously must be reviewed and approved by the PI as long as it is in remission.
9. Participation in another clinical study with an investigational product during the last 28 days.
10. Patients with documented cirrhosis (will need imaging +/- biopsy confirmation, hepatology consult recommended)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Measuring changes in dose limiting toxicities | Up to 28 days
  Determine the safety of adding Decitabine and Venetoclax to patients undergoing reduced intensity allogeneic transplantation for treatment of hematologic malignances with Fludarabine and Melphalan.

SECONDARY OUTCOMES:
The average regimen-related toxicity | At 1 year
  Rate of grade >- 4, non-hematologic toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Omer A Jamy, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States